CLINICAL TRIAL: NCT04507685
Title: Diet and Lifestyle Intervention Strategies to Treat β-cell Dysfunction and Insulin Resistance in Asian Indians
Brief Title: Asian Indian Prediabetes Study
Acronym: AIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: National Medical Research Foundation (NMRC) Singapore (Unknown); Almond Board of California (Other)
Responsible Party: Principal Investigator, Jeannie Tay, Senior Research Fellow, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-078
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pre Diabetes
Keywords: Asian Indians; Prediabetes; Insulin Resistance; Low glycaemic diet; Ectopic Fat
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State; Insulin Resistance | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: 24-week parallel arm, randomized controlled trial (RCT)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycaemic Diet (LG) (Experimental): Low carbohydrate, low saturated fat diet
  Interventions: Other: Lifestyle (Diet and Exercise)
- Control Diet (Active Comparator): High unrefined carbohydrate, low fat diet
  Interventions: Other: Lifestyle (Diet and Exercise)

INTERVENTIONS:
Other: Lifestyle (Diet and Exercise) — The LG diet will comprise 20% carbohydrate, 30% protein, and 50% fat (<10% saturated fat). It will have a low glycaemic load; include plant and animal protein; non-starchy vegetables and salad greens; and some low-sugar fruit. Participants will be encouraged to incorporate a variety of foods rich in monounsaturated and polyunsaturated fats in their diet.
  The control diet will comprise 50% carbohydrate, 20% protein and 30% total fat (<10% saturated fat). It will reflect the Health Promotion Board's (HPB) recommendations to reduce dietary fat, emphasize wholegrains and include a variety of fruits and vegetables. In contrast to the LG diet, the control diet will have a higher glycaemic load with a greater proportion of energy derived from unrefined carbohydrate foods.
  Concurrent to the dietary intervention and consistent with physical activity guidelines, all participants will undertake a 60-min structured exercise program incorporating aerobic/ resistance exercises 3-4 days/week.

SUMMARY:
Compared to other races, Indians have higher insulin resistance, poorer pancreatic function and a greater risk of developing diabetes, highlighting the importance of early strategies for improving insulin sensitivity and improving pancreatic function in Indians to prevent diabetes and lower the risk of heart disease.

A low carbohydrate diet can deplete fat from undesirable places, such as fat around organs in the abdominal cavity. In this study, we will determine if restriction of dietary carbohydrates will deplete fat in the pancreas and liver, and improve insulin sensitivity and early insulin secretion in Indians. These changes may prevent diabetes from developing. Hepatic and pancreatic fat will be measured using magnetic resonance imaging. Insulin sensitivity and secretion will be measured during an oral glucose tolerance test. In addition, this study will investigate if the higher insulin resistance in Indians is due to genes that cause the inability to store fat in the legs.

The results on the type of diet that is more effective for reducing pancreatic and hepatic fat is important for informing dietary guidelines on the use of low carbohydrate diets for diabetes prevention, particularly in Indians who have a higher risk of developing diabetes.

DETAILED DESCRIPTION:
Compared to other races, Indians have a greater risk of developing type 2 diabetes (T2D), increased insulin resistance (IR) and more rapid decline in β-cell function, highlighting the urgency and importance of early intervention strategies for improving insulin sensitivity and preserving/improving β-cell function to prevent T2D and mitigate against the increased vascular disease risk.

Preliminary findings show a reduction in glycemic load selectively depletes visceral and ectopic lipid and improves insulin sensitivity and β-cell function in non-diabetic adults. The proposed research will investigate if the phenotypic features increasing T2D risk in individuals of Indian ancestry (IR and impaired β-cell function) can be favorably modified by a low glycemic (LG) intervention, and if the increased IR is attributable to genetic factors regulating adipocyte differentiation and function.

These research objectives will be achieved through a 24-week randomized controlled trial (RCT) comparing isocaloric LG versus control diets in Indians with prediabetes. Compared to individuals in the control group, those on the LG diet are expected to have greater ectopic (pancreas, liver, visceral and intramyocellular) fat depletion assessed with MRI/MRS, and improvements in first phase insulin secretion and insulin sensitivity assessed with the C-peptide model and oral minimal model, respectively during an OGTT. Reductions in hepatic and pancreatic lipids will be associated with improvements in first-phase β-cell response. Individuals with a greater number of risk alleles from a 53-SNP IR genetic risk score will have lower insulin sensitivity and leg fat, supporting the notion that impaired adipocyte differentiation leading to limited peripheral adipose expansion capacity is an important etiological factor underpinning IR cardiometabolic disease in Indians.

The results will broaden the evidence base for effective prevention strategies in this high risk population by investigating the effect of the proposed diet intervention on underlying physiological and molecular mechanisms implicated in the pathophysiology of T2D in Indians.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Asian Indian ethnicity
* Age between 21-50 years
* BMI not greater than 35 or less than 25
* Prediabetes (based on results from an OGTT conducted in the last 3 months):

  * Impaired Fasting Glucose (IFG) which is a fasting blood glucose level of between 5.6 to 6.9 mmol/l and/or
  * Impaired Glucose Tolerance (IGT) which is a blood glucose level of 7.8 to 11.0 mmol/l, 2 hours after the OGTT but below 7.0 mmol/l in the fasting state.
* Not have type 1 or type 2 diabetes
* Not on any diabetes medications that affect insulin sensitivity e.g. metformin, glitazones
* No abnormality of clinical significance on medical history
* If female, not pregnant or breast feeding
* No history of coronary artery disease or cardiac (heart) abnormalities
* Participants must understand the procedures involved and agree to participate in the study by giving full informed, written consent

Exclusion Criteria:

* BMI greater than 35 or less than 25
* Weight gain or loss of more than 5% over the past 3 months
* Have anaemia (low haemoglobin/ red blood cell levels), a malignancy (cancer), abnormal liver function, any significant endocrinopathy (e.g. thyroid problems), or a history of metabolic disease such as liver, kidney, cardiovascular, respiratory or gastrointestinal disease.
* Have high uncontrolled hypertension (resting seated blood pressure >160/100 mmHg)
* Taking medications that may affect glucose metabolism e.g. steroids, thiazide diuretics at doses>25mg/day.
* History of smoking or using nicotine products during the 6 months prior to study
* History of heavy alcohol consumption (> 5 standard drinks/day)
* Inability to limit alcohol consumption for study duration
* Lactose Intolerant or have a nut allergy
* Have depression
* Have a musculoskeletal injury, joint or peripheral vascular disease sufficient to impede exercise (such as hip arthritis, foot, ankle problems or pain)
* Have severe exercise-induced asthma
* Participating in a regular aerobic or resistance exercise program
* Currently on a weight reducing diet or have an eating disorder
* Contraindications for MRI e.g. if you have certain metallic implants/devices such as heart valves of a cardiac pacemaker which may be affected by the magnetic field
* Unwilling to be randomized to either diet group
* Extended absences due to travel or other commitments
* Unable to comprehend or cope with study requirements

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in β-cell Function [First-phase β-cell response (PhiD)] | Week 0, 8 and 24
  First-phase β-cell response (PhiD) will be calculated from blood glucose and C-peptide data during a 3h 75g oral glucose tolerance test (OGTT) using the C-peptide minimal model.
Change in Insulinogenic index (ΔC-peptide/∆glucose during the first 30 minutes of the OGTT) | Week 0, 8 and 24
  ΔC-peptide/∆glucose during the first 30 minutes of the OGTT will be calculated as an index of early insulin secretion (Insulinogenic index).
Change in Incremental AUC | Week 0, 8 and 24
  Incremental AUC over 180 minutes of the OGTT will be calculated for glucose, insulin, and C-peptide.
Change in Insulin sensitivity (Oral Minimal model) | Week 0, 8 and 24
  Insulin sensitivity will be calculated from blood glucose, insulin and C-peptide during a 3h 75g oral glucose tolerance test (OGTT) using both the oral minimal model
Change in Matsuda index for whole body insulin sensitivity | Week 0, 8 and 24

SECONDARY OUTCOMES:
Change in Body fat distribution | Week 0, 8 and 24
  Body fat distribution will be imaged and quantified using MRI and MRS. Abdominal fat will be segmented to identify and quantify subcutaneous (deep and superficial) and visceral fat compartments. Lower body gluteal fat compartment will also be imaged and quantified. Fat within liver, pancreas and skeletal muscle fibers will be determined by MRI / MRS.
Change in Weight (kg) | Week 0, 8 and 24
Change in Blood Pressure | Week 0, 8 and 24
Change in Body Composition- Total body fat | Week 0, 8 and 24
  Total body fat (kg) will be assessed using DXA
Change in Body Composition- Total lean mass | Week 0, 8 and 24
  Total lean mass (kg) will be assessed using DXA
Genotyping analyses | Week 0
  Genomic DNA isolated from blood samples will be analysed
Change in Blood Lipids (total cholesterol, HDL-C, TAG, lipoprotein subfractions) | Week 0, 8 and 24
Change in liver enzymes | Week 0, 8 and 24
Change in inflammatory markers (e.g. IL-6, TNFα and CRP) | Week 0, 8 and 24
Change in satiety hormones (e.g. leptin, ghrelin, GIP and GLP-1). | Week 0, 8 and 24
Lipidomics | Week 0, 8 and 24
  Lipidomics evaluation of several lipid classes including sphingolipids (sphingomyelins, ceramides and glycosphingolipids) in plasma
Change in Plasma phospholipid fatty acid (FA) profile | Week 0, 8 and 24
Change in Gut microbiota composition | Week 0, 8 and 24
  Gut microbiota composition will be assessed by 16S or shotgun metagenomic sequencing
Change in Faecal characteristics- including short chain fatty acids (SCFAs). | Week 0, 8 and 24

OTHER OUTCOMES:
Change in respiratory quotient (RQ) | Week 0, 8 and 24
  Respiratory quotient (RQ) to assess substrate utilization by indirect calorimetry.
Change in blood ketone (β-hydroxybutyrate, βHB) concentrations | Week 0, 8 and 24
  A marker of carbohydrate intake
Change in 24-h urinary urea to creatinine ratio | Week 0, 8 and 24
  A marker of protein intake
Change in Physical activity levels | Week 0, 8 and 24
  Assessed with 7 consecutive days of triaxial accelerometry
Change in Exercise Classes attendance | 24 weeks
Change in dietary intake (diet checklists) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Tay, PhD, Principal Investigator — Institute for Human Development and Potential (IHDP), Singapore
Locations (1):
- Singapore Institute for Clinical Sciences (SICS), Singapore, Singapore